CLINICAL TRIAL: NCT00150293
Title: Pregabalin Open-Label Add-On Trial: An Open-Label, Multicenter Follow-On Study to Determine Long-Term Safety and Efficacy in Patients With Partial Seizures.
Brief Title: Evaluation of Long-Term Safety and Efficacy of Pregabalin in Patients With Partial Seizures.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1008-114
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Seizure Disorder, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Pregabalin

INTERVENTIONS:
Drug: Pregabalin

SUMMARY:
To determine long-term safety and efficacy of pregabalin in patients with partial seizures.

ELIGIBILITY:
Inclusion Criteria:

* Must have met the inclusion criteria for preceding double-blind study
* Have received double-blind study medication and wish to receive open-label pregabalin.

Exclusion Criteria:

* Cannot be pregnant or considering becoming pregnant during the course of the study.
* Cannot be receiving any concomitant medication that could alter the effectiveness of the pregabalin response or affect seizure frequency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337
Dates: Start 2002-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Safety Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (76):
- Australia (8):
  - Pfizer Investigational Site, Deakin, Australian Capital Territory
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Chastwood, New South Wales
  - Pfizer Investigational Site, Cairns, Queensland
  - Pfizer Investigational Site, Maroochydore, Queensland
  - Pfizer Investigational Site, Footscray, Victoria
  - Pfizer Investigational Site, Parkville, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
- Austria (5):
  - Pfizer Investigational Site, Auenbruggerplatz 22
  - Pfizer Investigational Site, Graz
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Vienna
- Pfizer Investigational Site, Leuven, Belgium
- Canada (14):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Penticton, British Columbia
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Barrie, Ontario
  - Pfizer Investigational Site, London, Ontario
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Windsor, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Québec, Quebec
  - Pfizer Investigational Site, Regina, Saskatchewan
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Germany (13):
  - Pfizer Investigational Site, Ulm, Baden-Wurttemberg
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bernau
  - Pfizer Investigational Site, Bonn
  - Pfizer Investigational Site, Dresden
  - Pfizer Investigational Site, Erlangen
  - Pfizer Investigational Site, Essen
  - Pfizer Investigational Site, Frankfurt
  - Pfizer Investigational Site, Freiburg im Breisgau
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Mainz
  - Pfizer Investigational Site, München
- Netherlands (3):
  - Pfizer Investigational Site, AE Breda
  - Pfizer Investigational Site, Blaricum
  - Pfizer Investigational Site, Ve Heeze
- Poland (14):
  - Pfizer Investigational Site, Bialystok
  - Pfizer Investigational Site, Bydgoszcz
  - Pfizer Investigational Site, Choroszcz
  - Pfizer Investigational Site, Gdansk
  - Pfizer Investigational Site, Grudziądz
  - Pfizer Investigational Site, Katowice
  - Pfizer Investigational Site, Krakow
  - Pfizer Investigational Site, Lublin
  - Pfizer Investigational Site, Mosina
  - Pfizer Investigational Site, Olsztyn
  - Pfizer Investigational Site, Poznan
  - Pfizer Investigational Site, Płock
  - Pfizer Investigational Site, Torun
  - Pfizer Investigational Site, Warsaw
- Portugal (2):
  - Pfizer Investigational Site, Coimbra
  - Pfizer Investigational Site, Porto
- Spain (6):
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Granada, Granada
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Zaragoza, Zaragoza
  - Pfizer Investigational Site, Girona
  - Pfizer Investigational Site, Madrid
- United Kingdom (9):
  - Pfizer Investigational Site, Middlesbrough, N. York
  - Pfizer Investigational Site, Washington, Tyne & Wear
  - Pfizer Investigational Site, Blackpool
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Leeds
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Northampton
  - Pfizer Investigational Site, Wolverhampton
- Pfizer Investigational Site